CLINICAL TRIAL: NCT05898698
Title: Prospective Observational Registry of Safety and Effectiveness of Acellular Fish Skin Grafts in Treatment of Cutaneous Wounds
Brief Title: Prospective Case Registry for Wounds
Status: Active, not recruiting | Type: Observational
Sponsor: Kerecis Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: KS-0790
Record Dates: First submitted 2023-06-01; First posted 2023-06-12 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-10

CONDITIONS: Wound Healing Delayed

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a post-market, observational and non-interventional registry to collect real-world data in diverse clinical settings and wound applications of acellular fish skin graft (FSG). The registry will be multi-center , target a wide patient population and a variety of wounds to document the quality of wound care, patient outcomes, safety and long-term results.

DETAILED DESCRIPTION:
Introduction: This registry will be conducted according to US standards of Good Clinical Practice as adopted by the Food and Drug Administration, associated Federal regulations and applicable institutional research policies and procedures. This study has been approved by a central IRB, WCG IRB in April 2023.

Registry Objectives: The overall objective of the registry is to collect quality and safety data to assess the efficacy of the FSG in treatment of acute and chronic wounds. The ultimate goal of the registry is to enhance quality of care, patient outcomes and establish a resource to facilitate the use of FSG in treatment of acute and chronic wounds.

Primary Objective: The main purpose of the registry is to evaluate the safety and long-term effectiveness of acellular fish skin grafts in treatment of acute and chronic wounds in a real world setting.

Secondary Objective: To evaluate the clinical and financial benefits of FSG in terms of quality of healing, pain and treatment cost.

Research Design: This registry will prospectively collect data from treatment and follow-up of patients who have undergone procedures where wounds are treated with Kerecis FSG. The registry is a non-experiment, multi-center , single arm, open label study to determine real world long-term safety and quality of Kerecis FSG. The study will not be interventional, de-indentified, HIPAA compliant data will only be collected on patients already scheduled to receive the Kerecis product. Subjects will be enrolled as they are scheduled to receive FSG for treatment of their index wound. Subjects will complete follow up as scheduled by their physician and their data will be documented at weekly follow-ups through week 32. Clinical improvement will be collected through case report forms (CRF) at each time point. Subjects will be followed for the 32 weeks but if the Index wound heals before that time , there will be a Healing Confirmation Visit (HCV) 2 weeks after to confirm the Index wound is still healed. If Index wound is not healed at the HCV then the subject will continue to next weekly visit. Index wound assessments will be captured digitally. The depth of the index wound will be collected manually by using a sterilized cotton swab placed in the deepest part of the wound and documenting that measurement. One year form the procedure, patients will receive a survey to evaluate their overall experience and provide any feedback. Overall, the registry is prospective except information regarding patient medical history can be collected retrospectively.

Registry Procedures: Specific Training: Prior to subject enrollment , the Sponsor will initiate in person training with participating sites to provide training to the physicians and their staff about the protocol, registry procedures and data entry. The sponsor will implement a number of strategies to ensure to ensure the quality, consistency and interpretability of data recorded. Training, education and ongoing liason with participating sites will be provided to support high quality data collection.

Data Management and Quality Plan: Data De-identification: Subjects enroll in the registry will be assigned a unique subject identification number. This number will consist of ten characters for the registry protocol number, three digits for a site number and four digits for a sequentially assigned subject number (i.e.,0001, 0002 etc.) Data confidentiality, storage, and Retention: All clinicians and related medical staff involved in looking after patients during the study are bound by medical confidentiality and are obliged to comply with data protection follow all Health Information Portability and Accountability Act of 1996 (HIPAA) and Protected Health Information (PHI). Data will be collected in a CRF and entered into secure, web-based portal databases. The databases are housed and managed in an International Organization for Standardization (ISO) 27001 certified environment. Only authorized users and site administrators can see site wide data. Surgeon users can only see their procedure. The registry will contain built-in exporting function to enable data extraction by participating sites to help clinicians review their practice and improve the services. The paper form CRF will be stored in a locked file cabinet at the participating sites and will be shredded after 7 years post completion of the registry.

Data Quality: The registry will implement several strategies to maintain data quality and consistency such as routine cleaning, quality check and periodic feedback. Training, education and ongoing liason with participating sites will be provided to supporting high quality data collection.

ELIGIBILITY:
Inclusion Criteria:

* Subjects age 18 and older and are able to provide informed consent.

Having at least one partial or full thickness wound appropriate for FSG and the wound has NOT received FSG previously.

Appropriate wounds include: Partial or full thickness wounds, Diabetic foot ulcers, venous leg ulcers, pressure ulcers, chronic vascular ulcers, Trauma wounds (2nd degree burn, abrasions, lacerations, skin tears.

Surgical wounds (donor sites/grafts, post-Mohs surgery, post Laser surgery, podiatric, wound dehiscence

Exclusion Criteria:

* Patient has a 3rd degree burn Patient has a know sensitivity to fish products Patient whose target wound was previously treated with FSG Patient is breastfeeding

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ages above 18 less than 90 years of age who have wounds being treated with FSG.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-03-17 (Actual); Primary Completion 2025-03-17 (Estimated); Study Completion 2025-12-17 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint : Complete Wound Closure | 32 weeks
  Is time and frequency of complete wound closure by or on 32 weeks. Complete closure is referred to as full epithelialization with the absence of drainage.

SECONDARY OUTCOMES:
Secondary Endpoints : Reduction in wound area | 32 weeks
  Proportion of subjects achieving > 60% reduction in wound area from baseline
Reduction in wound depth | 32 weeks
  Proportion of subjects achieving >60% reduction in wound depth from baseline
Increase in Vascularization | 32 weeks
  Proportion of subjects achieving >20% increase in revascularization ( or tissue oxygen saturation) from baseline using noninvasive imaging technique
Pain medication use | 32 weeks
  Proportion of subjects request for pain medication during treatment
Number of applications/Cost | 32 weeks
  Average number of FSG applications and average cost per patient until wound closes
Readmission rate | 32 weeks
  Number of readmission to hospital for index wound related event(s)
I year follow-up | 12 months
  12 month outcomes to see if any recurrences at the Index wound

CONTACTS AND LOCATIONS:
Locations (1):
- Kerecis, Arlington, Virginia, United States

IPD SHARING:
Plan to Share IPD: No